CLINICAL TRIAL: NCT00444158
Title: A Randomized, Double-Blind, Double-Dummy, 2-Period Crossover Study to Characterize the PK/PD Relationship of a 20-Minute Versus a 4-hour Intravenous Infusion of MOA-728 in Subjects on Stable Methadone Maintenance
Brief Title: Double-Blind, Double-Dummy, 2-Period Crossover of a 20-Minute Versus a 4-hour IV of MOA-728 in Stable Methadone Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3200L2-1108
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Constipation
Keywords: opioids; chronic pain
MeSH Terms: conditions — Constipation; Chronic Pain

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
MOA-728, an investigational drug, is currently being studied for the relief of constipation associated with postoperative ileus and treatment of opioid induced constipation in patients receiving palliative care. This study will further investigate the IV formulation of MOA-728 comparing PK/PD time points for a 20-minute versus a 4-hour infusion.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy men and nonlactating, nonpregnant women age 18 to 65 years with BMI of 18.0 to 35.0 kg/m2
* Must have been receiving methadone treatment of greater than or equal to 30 mg/day for at least one month and a positive drug screen for methadone
* High probability for compliance with and completion of the study

Exclusion Criteria:

* Significant cardiovascular, hepatic, renal , respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease. Presence or history of any disorder that may prevent the successful completion of the study. Any surgical or medical condition that my interfere with the distribution, metabolism or excretion of the test article.
* Acute disease state, family history of long QT syndrome and/or sudden cardiac death, allergy to opioids or drugs. Use of any investigational or prescription drugs within 30 days, any OTC drugs including herbal supplements within 14 days and drugs required to maintain regulation of bowel movements 48 hours before study day 1.
* History of alcoholism within 1 month before study day 1, admitted alcohol abuse, or consumption of more than 2 standard units of alcohol per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
It is not known if the activity of MOA-728 is related to the peak concentration or the overall exposure (AUC). This study is designed to evaluate the PK and PD effect of MOA-728 administered either as a 20-minute or 4-hour infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Gainesville, Florida, United States